CLINICAL TRIAL: NCT04188886
Title: Evaluation of the Daily Practices of ECMO Veino-arterial and Their Ethical Implications in France: Multicenter Observational Study (Evaluation of Professional Practice)
Brief Title: Evaluation of Practices of ECMO or ECLS and Ethical Implications in France
Acronym: EVAPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier La Chartreuse (Other)
Collaborators: Elodie BERG (Unknown)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, PI, Centre Hospitalier La Chartreuse
Other Study IDs: ElodieBERG2019
Record Dates: First submitted 2019-10-29; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Life Support Systems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Practice survey — Practice survey on

SUMMARY:
Short-term circulatory support (ECMO/ECLS) has become a common emergency resuscitation support.

Currently, the indication of the ECMO/ECLS relies more on clinic, biological and imagery arguments than on a real consensus.During the care of a patient under ECMO/ECLS, various stakeholders are involved in the implementation and its medical and paramedical management. Everyone, with their knowledge and experience, has an opinion on the relevance of this therapy.

DETAILED DESCRIPTION:
A validated questionnaire, translated from an Anglo-Saxon study, will be used as a basis for work and adapted. After the publication of a memo, it is accessible anonymously on a platform (ASKABOX) whose link is distributed by email by the secretaries or nursing staff. The city and the exercise service will be requested in the preamble of the questionnaire. It is composed of six demographic questions: age, gender, occupation, participation in emergency care, number of ECMOs encountered, level of knowledge about ECMO. The other questions concern concrete ECMO situations and the answers are nuanced from definitely yes to definitely no to allow professionals to express their opinion as well as possible. The targeted professionals are all those involved in the management of patients on ECMO: emergency physicians, anesthesiologists, surgeons, perfusionists, nurses, orderlies, ASHs.

A monocentric feasibility study was carried out with satisfactory results in terms of participation.

AN INFORMATION NOTE WILL BE ATTACHED WITH THE EMAIL AND THE LINK FOR THE QUESTIONNAIRE (ANONYMOUS)

ELIGIBILITY:
Inclusion Criteria:

* All medical and paramedical personnel involved in decision making, installation, and monitoring of the ECMO

Exclusion Criteria:

* MEDICAL AND PARAMEDICAL STAFF NOT INVOLVED IN THE ESTABLISHMENT OR FOLLOW-UP OF THE ECMO

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All medical and paramedical personnel involved in decision making, installation, and monitoring of the ECMO
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the involvement of professionals in ECMO-related decisions | 1 day
  Through an anonymous questionnaire, the investigators will evaluate the speciality (eg cardiac surgeon, anesthesiologist...) of the doctor responsible for the indication of ECLS

SECONDARY OUTCOMES:
Identification of the profession of each person involved in the management of the patients | 1 day
  Through an anonymous questionnaire, identifying the profession of each person involved in the management of the patients
Demographic data (age, sexe) of each personnel involved in the management of the patients | 1 day
  Through an anonymous questionnaire, identifying the demographic data of the health care staff involved in the care management of the patients
Level of training and knowledge of each personnel involved in the management of the patients | 1 day
  Through an anonymous questionnaire, identifying the level of training and knowledge of the health care staff involved in the care management of the patients
Opinion of the health care staff on the care management of the patients | 1 day
  Through an anonymous questionnaire, clarify the opinion of health care staff on care management

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bourgogne Franche Comté, Dijon, France

IPD SHARING:
Plan to Share IPD: No
The data will not be disclosed individually to other researchers. The analysis is done in a global way